CLINICAL TRIAL: NCT06922448
Title: A Phase 2a Randomized Double-blinded Placebo Controlled Study to Evaluate the Safety, Tolerability, PK, PD, and Preliminary Clinical Activity of BLU-808, a Wild-type KIT Inhibitor, in Participants With Ragweed (Ambrosia Artemisiifolia)-Induced Allergic Rhinoconjunctivitis
Brief Title: Study of BLU-808 in Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLU-808-2201
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergic Rhinoconjunctivitis; Ambrosia Artemisiifolia; BLU-808; Ragweed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BLU-808 Dose 1 (Experimental): BLU-808 will be administered orally for 28 days.
  Interventions: Drug: BLU-808
- BLU-808 Dose 2 (Experimental): BLU-808 will be administered orally for 28 days.
  Interventions: Drug: BLU-808
- Placebo (Placebo Comparator): Placebo will be administered orally for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLU-808 — BLU-808 tablets
  Arms: BLU-808 Dose 1; BLU-808 Dose 2
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of BLU-808 in participants with ragweed (Ambrosia artemisiifolia)-induced allergic rhinoconjunctivitis (ARC). Participants will undergo eligibility assessments that include exposure to ragweed pollen in an allergen exposure chamber (AEC).

ELIGIBILITY:
Key Inclusion Criteria

1. Adults, 18 years of age or older, willing to provide written informed consent, and willing to comply with all study requirements.
2. History (>2 years) of ragweed-induced ARC.
3. A positive ragweed skin prick test (mean diameter of ≥ 5 mm) in the last 6 months.
4. Must meet clinically relevant nasal and ocular symptoms as defined by the protocol.

Key Exclusion Criteria

Participants are excluded from the study if any of the following criteria are met:

1. Receiving medications (oral, nasal, topical, ocular, or injectable) to treat their ragweed or other allergy symptoms and/or receiving any medications that impact participants' safety or interfere with study assessments or interpretation of study results.
2. Have active rhinitis, sinusitis, and/or other severe allergies not associated with the ragweed pollen that may interfere with study symptom assessments.
3. Any prior or ongoing clinically significant illness, medical or psychiatric condition, surgical history, or physical finding that may interfere with the assessment or interpretation of study results.
4. Clinically significant moderate to severe, uncontrolled cardiovascular, renal or hepatic disease.
5. Significant bleeding risk or coagulation disorders.
6. Any form of smoking, vaping or history of alcohol and drug abuse.
7. Any malignancy within the past 5 years prior to Screening/AEC 1, except for basal cell or squamous cell carcinomas of the skin or carcinoma in situ.
8. Inadequately controlled asthma that could affect the safety of the participant or interfere with the assessment or interpretation of study results.
9. Known active/latent infection (viral, bacterial, fungal, helminth, or mycobacterial) such as tuberculosis, hepatitis B, hepatitis C, AIDS-related illness, or COVID-19 infection.
10. History of sinonasal conditions that may confound the assessment or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 through Day 56

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of BLU-808 | Day 1 to Day 28
Maximum Plasma Concentration (Cmax) of BLU-808 | Day 1 to Day 28
Minimum Plasma Concentration (Cmin) of BLU-808 | Day 1 to Day 28
Apparent Clearance (CL/F) of BLU-808 | Day 1 to Day 28
Apparent Volume of Distribution for the Central Compartment (Vc/F) of BLU-808 | Day 1 to Day 28
Terminal Half-life (t½) of BLU-808 | Day 1 to Day 28
Change in Baseline-adjusted Mean Total Nasal Symptom Score (TNSS) | Baseline, Day 14, Day 28
Change in Baseline-adjusted AUC of the TNSS | Baseline, Day 14, Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Red Maple Trials, Ottawa, Canada